CLINICAL TRIAL: NCT06271733
Title: Intensive PTSD Treatment Combined With Transcranial Magnetic Stimulation: A Randomized Controlled Study
Brief Title: TMS for Veterans Attending a 2-week Intensive Outpatient Program for PTSD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21110503
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active TMS (Active Comparator)
  Interventions: Device: TMS
- Sham (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: TMS — 2 sessions of iTBS per day for 5 days
  Arms: Active TMS
Device: Sham — 2 sessions per day for 5 days of sham condition
  Arms: Sham

SUMMARY:
The goal of this study is to determine whether complementing regular intensive PTSD treatment with intermittent theta burst stimulation (iTBS) applied to the right dorsolateral prefrontal cortex (DLPFC) can improve treatment response for individuals attending a 2-week intensive outpatient program (IOP) for PTSD. Specifically, the present study will compare iTBS versus a sham condition during the second week of the 2- week IOP for veterans who have not experienced PTSD symptom reductions over the course of the first week of the Road Home Program intensive PTSD treatment program.

DETAILED DESCRIPTION:
Despite the efficacy of many evidence-based treatments for psychiatric disorders, a large percentage of treatment completers maintain their diagnosis and symptoms after treatment. For veterans with PTSD, approximately 66% of all individuals who successfully complete an evidence-based treatment retain their PTSD diagnosis.

An intervention that has been shown to be effective for non-response to first-line psychotherapies is transcranial magnetic stimulation (TMS). TMS is a safe, noninvasive intervention that uses a magnetic field to modulate cortical activity in brain areas linked to an overactive stress response. When compared to sham conditions which resembles the TMS condition but does not utilize any magnetic fields (i.e., proposed active ingredient), TMS has been associated with reduced depressive symptoms in treatment non-responders. Although the bulk of research examines TMS as a treatment for major depressive disorder, TMS has also shown promise in reducing symptoms of other psychiatric disorders such as PTSD.

In prior research TMS was associated with medium to large reductions in core PTSD symptoms when compared to sham conditions. Symptom reductions achieved via TMS have been demonstrated to persist. A recent study compared Cognitive Processing Therapy (CPT) combined with TMS to CPT with a sham condition and found that CPT combined with TMS was associated with greater PTSD symptom reductions during treatment and at six-month follow-up than CPT combined with a sham condition. This finding suggests that TMS may be beneficial as an augmentation to CPT. However, to our knowledge, previous literature has not yet examined whether TMS improves outcomes for individuals who are likely to not respond to CPT treatment.

Due to the demand for briefer TMS protocols, theta burst stimulation (iTBS) is a variation on TMS. Studies have found iTBS to be more efficient than standard TMS but still associated with significant improvements and low side effects in both depression and PTSD. The present study will utilize the more efficient iTBS protocol applied to the right dorsolateral prefrontal cortex (DLPFC) in order to reduce the length of stay for the participants.

Roughly one in four participants who complete Cognitive Processing Therapy (CPT) in the 2-week intensive outpatient program (IOP) at the Road Home Program at Rush do not report a meaningful reduction in PTSD symptoms and can be classified as non-responders. The present study seeks to determine whether adding iTBS to standard IOP programming reduces PTSD symptoms to a greater extent than adding a sham condition among participants who have not reported reduced symptoms by the end of the first week of treatment (i.e., likely non-responders). The present study will compare the two conditions at both post-treatment, 1- and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Veterans or service members between the ages of 18 and 65 who are attending the 2- week Intensive Outpatient Program at the Road Home Program and have not had significant PTSD symptom change based on the PCL-5 during the first week of treatment.
* Participants with an HDRS-21 score ≤ 26 at screening visit

Exclusion Criteria:

* Individuals with implants and non-removable metals which prevent them from safely receiving TMS, including:

  * Aneurysm clips or coils
  * Stents in the head, neck, or brain
  * Deep brain stimulators
  * Metallic implants in the head, neck, or brain (braces and dental implants do not interfere and are safe for TMS)
  * Shrapnel or bullet fragments in or near the head
  * Facial tattoos with metallic or magnetic-sensitive ink
  * Other metal devices or ferromagnetic objects implanted in or near the head
  * Pacemakers, intra-cardiac lines, or implanted medical pumps
* Individuals with a history of seizures or epilepsy (except those therapeutically induced by ECT)
* Individuals diagnosed with major, chronic mental health illnesses such as Psychotic Disorders, Bipolar Disorders, and Obsessive Compulsive Disorder
* Individuals with a history of substance abuse within the past six months
* Individuals with significant neurological disorders such as Parkinson's disease, Huntington's chorea, and Multiple sclerosis
* Individuals with unstable physical disease, such as unstable cardiac diseases
* Individuals currently on Benzodiazepine at a dose higher than 3mg or Lorazepam or equivalent.
* Women who are breastfeeding or pregnant
* Individuals with previous TMS treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Baseline, 1 month follow up
  Measure of PTSD symptom severity

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 1 month follow up
  Measure of depression symptom severity

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No